CLINICAL TRIAL: NCT03103529
Title: Safety and Feasibility of Early Active Rehabilitation in Children After Concussion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Isabelle Gagnon, Clinician Scientist/Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-142-PED
Record Dates: First submitted 2017-04-01; First posted 2017-04-06 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Post-Concussion Symptoms; Concussion
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Rehab (Experimental): Children will begin active rehabilitation 2 weeks post-injury
  Interventions: Other: Active Rehabilitation
- late rehab (Active Comparator): Children will begin active rehabilitation 4 weeks post-injury
  Interventions: Other: Active Rehabilitation

INTERVENTIONS:
Other: Active Rehabilitation

SUMMARY:
It has been suggested that activity immediately following concussion is detrimental to recovery and may lead to long term impairments. The animal model has shown that exercise too soon can lead to neurometabolic energy imbalances within the brain. However, there is also evidence to suggest that prolonged inactivity has negative consequences that may contribute to prolongation of symptoms. Determining the ideal timeframe in which to initiate an active rehabilitation protocol for patients who are slow to recovery is an important factor in concussion management.

ELIGIBILITY:
Inclusion Criteria:

* referred to the mTBI clinic of the MCH for atypical recovery (defined as the presence of symptoms with little improvement at 10 days post-injury preventing them from entering standard return to activities protocols)

Exclusion Criteria:

* co-morbidity preventing children from participating in intervention

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Post-concussion symptoms | 6 weeks post-injury
  Post-Concussion Symptoms Inventory scale total score

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Children's Hospital, MUHC, Montreal, Quebec, Canada